CLINICAL TRIAL: NCT06196866
Title: Effectiveness of Two Different Exergaming Systems in Addition to Conventional Treatment for Physical Therapy in Patients with Multiple Sclerosis: a Study Protocol for a Multicenter, Assessor-blind, 24-week, Randomized Controlled Trial
Brief Title: Effectiveness of Exergaming in Adittion to Conventional Treatment for Physical Therapy in People with Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Alvaro Alba Rueda, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESCMU01
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Exergaming; Nintendo Wii Fit; Nintendo Ring Fit Adventure; Physical therapy; Randomized controlled trial; Neurological rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): Participants carry out daily routine activities and/or receive standard physiotherapy for the whole 24 weeks of the trial, 1 session/week with a time of 45 minutes/session.
  Interventions: Other: Conventional Therapy
- Exergaming group 1 (Experimental): Participants receive Nintendo Ring Fit Adventure exergaming intervention for 12 weeks, 1 session/week with a time of 45 minutes/session + Control group intervention.
  Interventions: Device: Nintendo Ring Fit Adventure + Conventional Therapy
- Exergaming group 2 (Experimental): Participants receive Nintendo Wii Fit exergaming intervention for 12 weeks, 1 session/week with a time of 45 minutes/session + Control group intervention.
  Interventions: Device: Nintendo Wii Fit + Conventional Therapy

INTERVENTIONS:
Other: Conventional Therapy — The control group will develop only conventional treatment for the whole trial (weeks 1-24), consisting of carrying out daily routine activities and/or 1 session/week of physiotherapy (which includes manual therapy, active exercises of repetition of functional movements, walking, stairs and stretching) with a time of 45 minutes/session.
  Arms: Control group
Device: Nintendo Ring Fit Adventure + Conventional Therapy — In the exergaming group 1, the intervention will be 12 weeks (weeks 1-12) with a frequency of 1 session/week and with a time of 45 minutes/session, in addition to the users' conventional therapy. The training will be a first 5 minutes warm-up (composed of joint mobility and global stretching), 35 min of exergaming training (working on the participants' gait, stability and global muscle strength) and last 5 minutes of cooling down (composed of breathing exercises, joint mobility and global stretching) in each session. The therapist will choose in each session different exercises from each of these 4 sections:
  Jogging: Begginia or Transient Temple.
  Minigames: Squat Goals, Squattery Wheel, Gluting Gallery, Thigh Rider, Bank Balance or Dreadmill.
  Lower Limbs Training: Knee Lift or Hip Lift.
  Yoga: Tree Pose or Chair Pose.
  Arms: Exergaming group 1
Device: Nintendo Wii Fit + Conventional Therapy — In the exergaming group 2, the intervention will be 12 weeks (weeks 1-12) with a frequency of 1 session/week and with a time of 45 minutes/session, in addition to the users' conventional therapy. The training will be a first 5 minutes warm-up (composed of joint mobility and global stretching), 35 min of exergaming training (working on the participants' gait, stability and global muscle strength) and last 5 minutes of cooling down (composed of breathing exercises, joint mobility and global stretching) in each session. The therapist will choose in each session different exercises from each of these 4 sections:
  Aerobics: Basic Run or Hula Hoop.
  Strength Training: Rowing Squat, Single-Leg Extension, Sideways Leg Lift or Single-Leg Twist.
  Balance Games: Ski Jump, Balance Bubble, Table Tilt or Penguin Slide.
  Yoga: Chair or Standing Knee.
  Arms: Exergaming group 2

SUMMARY:
The present study aims to evaluate the effectiveness of two different exergaming systems in addition to conventional treatment on physical functional capacity, balance, muscle strength, spasticity in lower limbs and quality of life compared to an isolated conventional intervention in patients with multiple sclerosis. The secondary aim will be to compare the differences between both exergaming groups.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic autoimmune inflammatory disease of the central nervous system, which produces demyelination and axonal damage in the brain and spinal cord. Since there is currently no treatment for this condition, the goal of rehabilitation is to assist people with their manifestations. Over the last decade, exergaming with commercial consoles has demonstrated potential benefits in managing motor and functional impairments. However, new videogame strategies and assessment in randomized controlled trials are necessary to obtain significant results in different outcomes.

The hypothesis is that the exergaming systems in addition to conventional treatment will show statistically significant improvements on motor skills, spasticity, and quality of life results compared to conventional therapy alone. Therefore, this project aims to evaluate the effectiveness of two different exergaming systems in addition to conventional treatment on physical functional capacity, balance, muscle strength, spasticity in lower limbs and quality of life compared to an isolated conventional intervention in patients with multiple sclerosis. The investigators here design a multi-center, assessor-blind, 24-weeks, randomized controlled trial protocol. The achievement of the present project would serve to analyze the benefits of an alternative exercise program in the motor and functional rehabilitation program of multiple sclerosis patients and to identify the subjects in whom the benefits would be greater and whose implementation would have greater priority.

ELIGIBILITY:
Inclusion Criteria:

(i) Diagnosis of MS in any of its types (clinically isolated syndrome, relapsing-remitting MS, primary progressive MS or secondary progressive MS) based on the McDonald criteria.

(ii) Age over 18 years.

(iii) Mini-Mental State Examination score > 19 points.

(iv) Score on the Expanded Disability Status Scale (EDSS) under 7.0 points.

Exclusion Criteria:

(i) Diagnosis of another disease that affects balance and/or coordination.

(ii) Exacerbation or steroid treatment in the 30 days prior to inclusion in the study.

(iii) Presence of visual deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Physical Functional Capacity (6MWT) | Initial baseline assessment (week 1), assessment post-intervention 1 (week 12) and assessment post-intervention 2 (week 24).
  Physical functional capacity will be measured by 6-minute walk test (6MWT), a stress test that measures the maximum distance that an individual can travel during a period of six minutes walking as fast as possible. It will be carried out in a corridor 30 meters long, with a flat surface, preferably indoors and avoiding the traffic of people not involved in the test. Heart rate and O2 saturation (using a pulse oximeter) at the beginning and end of the test and the Borg scale (perception of effort) will also be compared.
Quality Of Life (MSQOL-54) | Initial baseline assessment (week 1), assessment post-intervention 1 (week 12) and assessment post-intervention 2 (week 24).
  The quality of life will be measured by the Multiple Sclerosis Specific Quality of Life Questionnaire (MSQOL-54). This questionnaire consists of 54 items distributed in 12 scales that measure the following dimensions of quality of life: physical health, limitations due to physical problems, limitations due to emotional problems, pain, emotional well-being, energy, health perception, social function, cognitive function, health concern, overall quality of life, sexual function, changes in health, satisfaction with sexual function. It was created from the SF-36, completing it with 18 additional items on specific aspects of multiple sclerosis.
Balance (Tinetti Balance Scale) | Initial baseline assessment (week 1), assessment post-intervention 1 (week 12) and assessment post-intervention 2 (week 24).
  The balance will be measured by the Tinetti Balance Scale. The scale qualifies the subject's static and dynamic balance during walking through 16 items, thus early detecting the risk of suffering a fall. The maximum score for static balance is 16 points and for balance during walking is 12 points, with the total sum of the scale being 28 points. It is considered a high risk of falls: less than 19 points; moderate risk of falls: from 19 to 23 points, and low or mild risk: from 24 to 28 points.
Strength in Lower Limbs (Handheld dynamometer) | Initial baseline assessment (week 1), assessment post-intervention 1 (week 12) and assessment post-intervention 2 (week 24).
  The strength in the lower limbs will be measured by a handheld dynamometer (HHD). The instrument for measuring the maximum isometric voluntary contraction of the muscles will be involved in the different joint movements. The protocol will consist of two consecutive maximum contractions for each muscle group, preceded by a warm-up test. Participants will first be shown the movement to be performed and then asked to perform it to confirm their understanding and begin the warm-up. The two measurements will be carried out continuously for 6 seconds with intervals of 30 seconds between contractions for greater performance. The final value will be the average of the two measurements made. The measurements will be carried out on the dominant lower limb in hip flexors, hip extensors, hip adductors, hip abductors, knee flexors, knee extensors, ankle flexors and ankle extensors muscles.
Spasticity in Lower Limbs (Modified Ashworth Scale) | Initial baseline assessment (week 1), assessment post-intervention 1 (week 12) and assessment post-intervention 2 (week 24).
  The spasticity in the lower limbs will be measured by Modified Ashworth Scale (MAS). This clinical tool will be used to assess muscle tone by measuring the level of resistance to passive movement. Compared to the original version, this scale includes the score 1+, thus existing a range between 0 (no increase in tone) and 4 (affected part rigid in flexion or extension) with 6 different options. These passive joint movements will be performed between 5-8 times (for a more reliable result) in 1 second from the position of maximum contraction of the muscle to be evaluated. The protocol will consist of carrying out the evaluation on a stretcher after 3 minutes of rest on it (thus avoiding the possible increase of muscle tone due to movement). Passive movements will be carried out in both lower limbs (starting with the left leg) in hip flexors, hip extensors, hip adductors, hip abductors, knee flexors, knee extensors, ankle flexors and ankle extensors muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Amaranta De Miguel Rubio, PhD, Study Director — Universidad de Córdoba; David Lucena Anton, PhD, Study Director — University of Cadiz
Locations (1):
- University of Cordoba, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No